CLINICAL TRIAL: NCT00532506
Title: Phase II Dose-Finding Study of SK-0403 With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DP1001
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: SK-0403

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of SK-0403 in patients with Type2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive subjects diagnosed with type 2 diabetes mellitus
* Stable diet program for at least 8 weeks
* Criteria for HbA1c are met

Exclusion Criteria:

* Type 1 diabetes
* Patients treated with other antidiabetic drugs or Insulin

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ryuzo Kawamori, M.D., Study Chair — Juntendo University School of Medicine, Dept. of Endocrinology and Metabolism
Locations (10):
- Japan (10):
  - Fukuoka
  - Gifu
  - Gunma
  - Hokkaido
  - Ibaraki
  - Kanagawa
  - Kumamoto
  - Okinawa
  - Ōita
  - Tokyo